CLINICAL TRIAL: NCT00581425
Title: Intron-A/Aldara Combination Therapy for BCC Excluding the Face and Scalp
Brief Title: Intron-A/Aldara Combination Therapy for Basal Cell Carcinoma (BCC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Stephen Tucker, Visiting Professor - Dermatology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-06-0478; OSP-24412
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Basal Cell Carcinoma
Keywords: BCC; Basal Cell Carcinoma; Intron-A; Aldara; Basal Cell Carcinoma excluding scalp and face
MeSH Terms: conditions — Carcinoma, Basal Cell; Facies | interventions — Imiquimod; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated (Experimental)
  Interventions: Biological: Imiquimod and Interferon alpha

INTERVENTIONS:
Biological: Imiquimod and Interferon alpha — Imiquimod first two weeks and last two weeks. Interferon middle five weeks.

SUMMARY:
A trial to see if BCC excluding the scalp and face can be treated successfully with a combination therapy of Intron-A and Aldara.

ELIGIBILITY:
Inclusion Criteria:

* Nodular or superficial basal cell carcinoma on the skin excluding scalp or face

Exclusion Criteria:

* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
resolution of basal cell carcinoma | 2 years

SECONDARY OUTCOMES:
resolution of basal cell carcinoma at a lower cost and less inflammation. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Tucker, M.D., Principal Investigator — University of Texas Health Science Center of Houston Dermatology Clinic
Locations (1):
- University of Texas Health Science Center of Houston Dermatology Clinic, Houston, Texas, United States